CLINICAL TRIAL: NCT01214369
Title: Anesthetic Efficacy of X-tip Intraosseous Injection Following Mandibular Nerve Block in Molars With Acute Irreversible Pulpitis
Brief Title: Anesthetic Efficacy of X-tip Intraosseous Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Professor Mohammad Ramezani, Faculty of pharmacy, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 88288
Record Dates: First submitted 2010-09-10; First posted 2010-10-05 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-09

CONDITIONS: Anesthesia
Keywords: intraosseous injection; X-tip; PDL injection; Supplementary Injection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- X-tip intraosseous injection (Active Comparator)
  Interventions: Procedure: Type of Supplementary Injection
- PDL injection (Active Comparator)
  Interventions: Procedure: Type of Supplementary Injection

INTERVENTIONS:
Procedure: Type of Supplementary Injection — Patients will be selected from a group who were not anesthetized following 3.6 ml block injection. Half of the randomly selected patients will receive X-tip intraosseous injection and half will receive PDL injection as a supplementary for completing the anesthesia in selected hot mandibular molar teeth.

SUMMARY:
* Hypothesis:

  * X-tip intraosseous is an effective supplementary injection in mandibular hot teeth as well as Periodontal Ligament (PDL) injection
* Purposes:

  * Comparing the anesthetic efficacy of X-tip intraosseous and PDL injection in mandibular hot teeth which had not been anesthetized after 3.6 ml Infra Alveolar Nerve Block
* Methods and Materials:

  * forty patients with mandibular hot molar or second premolar which had not been anesthetized after 3.6 ml inferior alveolar nerve block injection will be selected for this study

DETAILED DESCRIPTION:
* Randomization:

  * All patients will be randomly divided into two groups as follows:

    1. X-tip intraosseous injection will be used as supplementary
    2. PDL injection will be used as supplementary
* Anesthetic evaluation:

  * For anesthetic evaluation we will use Visual Analog Scale (VAS)

ELIGIBILITY:
Inclusion Criteria:

* Mandibular Molars and second premolars with Acute Irreversible Pulpitis
* None of the teeth selected should have been anesthetized following 3.6 ml Lidocaine block injection

Exclusion Criteria:

* Unhealthy patients
* Teeth which were anesthetized following 3.6 ml nerve block injection
* Patients who did not have any signs of lip anesthesia following 3.6 ml injection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-11 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Number of participant who will have the pain following X-tip or PDL as a supplementary injection | 6 months
  All particiapant will be asked to show their pain degree on VAS for evaluation the efficacy of injections as a supplementary for anesthetising the teeth before and after the supplementary injection.

SECONDARY OUTCOMES:
Heart rate monitoring | before block injection and after supplementary injection
  This record will be monitored by puls oximeter device

CONTACTS AND LOCATIONS:
Overall Officials: Jamileh Ghoddusi, DDS,MSc, Principal Investigator — Dental Research Center,Faculty of Dentistry, Mashhad University of Medical Sciences, Iran
Locations (1):
- Faculty of Dentistry, Mashhad, Khorasan Razavi, Iran